CLINICAL TRIAL: NCT06758349
Title: OPErA Orchestral Posture Egonomic Assessment
Acronym: OPErA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: 09_16/12/2022
Record Dates: First submitted 2024-07-12; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Abnormal Posture
Keywords: Abnormal posture; Musician; Pain; functional limitation
MeSH Terms: conditions — Pain | interventions — Sitting Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orchestral musicians: The enrolled sample will consist of 250 professional musicians from major Italian orchestras.
  Interventions: Other: General questionnaire; Other: Pain Questionnaire; Other: Postural assessment without musical instrument in sitting position; Other: Postural assessment with the instrument in sitting position.

INTERVENTIONS:
Other: General questionnaire — Demographic, medical history, and musical activity data will be collected using a specifically designed questionnaire
Other: Pain Questionnaire — Questionnaire that evaluate pain and functional limitation during last week, last six months e during the carrier.
  The impact of painful symptoms on professional and non-professional activities , during the last week, will be assessed using the QuickDASH scale for the upper limb, the Modified Oswestry Low Back Disability Index for low back pain, and the Neck Disability Index questionnaire for cervico-dorsalgia
Other: Postural assessment without musical instrument in sitting position — Postural assessment without the instrument in a sitting position. Disposable ECG electrodes will be applied to the following anatomical landmarks: Spinous process C7 (C7), Right shoulder acromion (RS), Left shoulder acromion (LS), Right scapula inferior angle (RIA), Left scapula inferior angle (LIA), Spinous process L3 (L3), Intergluteal line (IG), vertex. The Physical Analyzer Portable will be used: a non-invasive, portable device that allows calibrated photo acquisition on the frontal and sagittal planes and subsequent data processing through dedicated software. On frontal plane they will be calculated: Trunk inclination, Head-neck inclination, Right and left shoulder height, Right and left shoulder width, right and left scapula-rachis distance. On sagittal plane they will be calculated: cervical and lumbar arrow, right and left shoulder distance.
Other: Postural assessment with the instrument in sitting position. — Postural assessment with the instrument in a sitting position. Disposable ECG electrodes will be applied to the following anatomical landmarks: Spinous process C7 (C7), Right shoulder acromion (RS), Left shoulder acromion (LS), Right scapula inferior angle (RIA), Left scapula inferior angle (LIA), Spinous process L3 (L3), Intergluteal line (IG), vertex. The Physical Analyzer Portable will be used: a non-invasive, portable device that allows calibrated photo acquisition on the frontal and sagittal planes and subsequent data processing through dedicated software. On frontal plane they will be calculated: Trunk inclination, Head-neck inclination, Right and left shoulder height, Right and left shoulder width, right and left scapula-rachis distance. On sagittal plane they will be calculated: cervical and lumbar arrow, right and left shoulder distance.

SUMMARY:
This is an observational study that will allow to understand if and how posture at the instrument can affect musician health and ability to work.

The study will last 3 years during which the investigators will evaluate 250 orchestral players: all musical instruments will be included. Postural assessments will be performed in the various venues of the participating orchestras.

The study participant, would initially answer a questionnaire that will investigate lifestyle habits (physical activity), professional activity (e.g. instrument played, hours of study/work, study methods) and general health (e.g. presence of pain with functional limitation at the present time or in the past, diagnosis of scoliosis).

The subsequent postural assessment will consist of two phases: phase 1 without an instrument in a sitting position, phase 2 with the musical instrument .

Disposable ECG electrodes will be applied to the skin and will serve as landmarks and will be removed at the end of the assessment.

In both phases, the Physical Analyzer Portable system will be used, which allows the acquisition of calibrated photographs and the subsequent processing of the data obtained through special software, calculating with numerical values the postural asymmetries between the right and left sides and the degrees of inclination of the trunk.

The execution of the planned assessments will take place in the constant presence and under the guidance and control of suitable and qualified personnel who will provide instructions on the activity to be carried out and assistance in case of any need.

The data obtained in this way will be correlated with the information collected with the questionnaire.

Improving musician posture awareness with the musical instrument could prevent the onset of pain and limitations in work activity.

In fact, the identification of risk factors for musculoskeletal pathologies in professional musicians (PRMDs) would allow the development of specific prevention and treatment programs and the development of a network of territorial services dedicated to the musicians themselves.

DETAILED DESCRIPTION:
For musicians, movement takes on a particular significance as it allows them to express their creativity through their instrument. The sensation they convey to the audience is one of a body in perfect harmony and symbiosis with their instrument, seemingly free of muscular tension and pain. However, numerous musculoskeletal and neurological disorders afflict musicians, limiting their performance and sometimes forcing them to cease their professional activity. Musicians often tend to underestimate their problems, ignoring pain and symptoms that require care or rest.

In 1713, Bernardino Ramazzini was the first to describe an overview of occupational diseases affecting musicians. Zaza, on the other hand, was the first to introduce the term Playing-Related Musculoskeletal Disorder (PRMD) to define musculoskeletal afflictions as "chronic, disabling personal health problems that affect the entire person physically, emotionally, and in terms of work and social aspects".

Recent systematic reviews report a prevalence of musculoskeletal disorders among musicians ranging from 57% to 68%, PRMDs from 9% to 68%, and one-time PRMDs from 62% to 93%. Fishbein highlighted that approximately 76% of members of the International Conference of Symphony and Opera Musicians (ICSOM) experienced at least one medical issue in their career that compromised their performance.

To find effective solutions for preventing the development of PRMDs or minimizing their impact, it is essential to first identify the main risk factors. The most frequently cited factors in the development of PRMDs include gender, age, professional status and years of experience, type of instrument, repertoire, individual technique, long hours of practice with insufficient breaks, poor physical condition, muscle fatigue, lack of preventive behaviours, and previous injuries. Additionally, several studies have revealed a correlation between the presence of musculoskeletal disorders and psychological stress factors (anxiety and stress, depression, and perfectionism). The weight of the instrument and the imposed posture may also influence the prevalence of musculoskeletal injuries among musicians.

Many researchers confirm that prolonged adoption of forced body positions required to play a specific instrument increases the likelihood of overloading the osteo-artro-neuromuscular system. However, few researchers have attempted to clarify the influence of playing classical musical instruments on posture. On average, a musician plays 1300 hours per year in an ergonomically unfavourable position. Instruments that require different positions and playing techniques are associated with varying prevalence of musculoskeletal disorders. A study conducted among conservatory students highlighted a high prevalence of postural alterations without the instrument (66.2%) and a non-optimal posture with the instrument in 73.4% of cases. Instruments that impose asymmetrical postures, such as the violin, viola, and flute, were found to be the main risk factors for incongruent postures.

Musicians who play with their arms above the scapulo-humeral plane are also more prone to suffer from PRMDs in the upper limb compared to those who play in a neutral position. Correcting these conditions, which represent one of the main risk factors for the development of musculoskeletal disorders in workers, depends on understanding the influencing factors and implementing an appropriate therapeutic and preventive approach.

Regarding the ergonomic risk assessment in orchestra musicians, recent reviews have highlighted that there are few publications on this subject. There is more information available on questionnaires used to assess symptoms reported by musicians due to inflammatory processes and musculoskeletal disorders, such as the "Standardized Nordic Questionnaire"; the DASH (Disabilities of the Arm, Shoulder, and Hand), and the MPIIQM (Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians).

The objectives of the study on a sample of orchestra musicians are:

* To study the prevalence of abnormal posture with and without instruments and describe them quantitatively.
* To investigate whether and which abnormal posture are associated with pain and PRMDs.
* To identify any risk factors for the development of abnormal posture, pain, and PRMDs.
* To study the impact of abnormal posture and PRMDs on professional life. If the study hypothesis is confirmed, it would demonstrate the high prevalence of abnormal posture among professional musicians and the significant impact on their performance and professional activity. Another effect would be raising awareness among professional musicians about the physical stresses they are exposed to and the disorders they may develop, which are still often misunderstood and underestimated by the musicians themselves.

Confirming our hypothesis would concurrently lead to an enhancement of the ongoing activities.

ELIGIBILITY:
Inclusion Criteria:

* Professional musicians from major Italian orchestras

Exclusion Criteria:

- Pain associated with acute trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: orchestral musicians playing symmetrical and asymmetrical musical instruments
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Pain, Limitation and Posture last week | the week prior to the assessment
  The investigators will evaluate if there is a correlation between pain with and without functional limitation with the following measure: trunk inclination, cervical inclination, dorsal curve, lumbar curve , right shoulder position, right shoulder height, right scapulae, left shoulder position, left shoulder height, left scapulae last week before the assessment
Pain, Limitation and Posture last six months | the six months prior to the assessment
  The investigators will evaluate if there is a correlation between pain with and without functional limitation with the following measure: trunk inclination, cervical inclination, dorsal curve, lumbar curve , right shoulder position, right shoulder height, right scapulae, left shoulder position, left shoulder height, left scapulae during the last 6 months before the assessment

SECONDARY OUTCOMES:
Prevalance of pain without functional limitation during last week | the week prior to the assessment
  The investigators will calculate the prevalance of pain without functional limitation for the week prior to the assessment using questionnaire data
Prevalence of pain without functional limitation during last six months | the six months prior to the assessment
  The investigators will calculate the prevalance of pain without functional limitation for the six months prior to the assessment using questionnaire data.
Prevalance of pain with functional limitation during last week | the week prior to the assessment
  The investigators will calculate the prevalance of pain with functional limitation for the week prior to the assessment using questionnaire data
Prevalence of pain with functional limitation during last six months | the six months prior to the assessment
  The investigators will calculate the prevalance of pain with functional limitation for the six months prior to the assessment using questionnaire data.
Pain with o without functional limitation during last week and personal and playing habit | the week prior to the assessment
  The investigators will evaluate if there is a correlation between the "prevalance of pain with and without functional limitation during last week" with the personal and playing habits collected with the questionnaire.
Pain with o without functional limitation during last six months week and personal and playing habit | the six months prior to the assessment
  The investigators will evaluate if there is a correlation between the "prevalance of pain with and without functional limitation during last six months" with the personal and playing habits collected with the questionnaire.
Degrees of Trunk Rotation (TR) | at the assessment time
  The investigators will calculate in degrees the difference between trunk rotation with and without musical instrument measured by the Physical Analyzer Portable .
Degrees of Trunk Inclination (TI) | at the assessment time
  The investigators will calculate in degrees the difference between trunk inclination with and without musical instrument measured by the Physical Analyzer Portable .
Degrees of Cervical Inclination (CI) | at the assessment time
  The investigators will calculate in degrees the difference between cervical inclination with and without musical instrument measured by the Physical Analyzer Portable .
Right shoulder vertical shift | at the assessment time
  The investigators will calculate in millimeters the difference between right shoulder height with and without musical instrument measured by the Physical Analyzer Portable .
Left shoulder vertical shift | at the assessment time
  The investigators will calculate in millimeters the difference between left shoulder height with and without musical instrument measured by the Physical Analyzer Portable .
Right shoulder sagittal shift | at the assessment time
  The investigators will calculate in millimeters the difference between right shoulder position on sagittal plane with and without musical instrument measured by the Physical Analyzer Portable .
Left shoulder sagittal shift | at the assessment time
  The investigators will calculate in millimeters the difference between left shoulder position on sagittal plane with and without musical instrument measured by the Physical Analyzer Portable .
Right Scapula lateral shift | at the assessment time
  The investigators will calculate in millimeters the difference between right scapula position with and without musical instrument measured by the Physical Analyzer Portable .
Left scapula lateral shift | at the assessment time
  The investigators will calculate in millimeters the difference between left scapula position with and without musical instrument measured by the Physical Analyzer Portable .
Dorsal curve change | at the assessment time
  The investigators will calculate in millimeters the difference between dorsal curve with and without musical instrument measured by the Physical Analyzer Portable .
Lumbar curve change | at the assessment time
  The investigators will calculate in millimeters the difference between lombar curve with and without musical instrument measured by the Physical Analyzer Portable .

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Santa Maria Nascente Fondazione Don Carlo Gnocchi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramella M, Fronte F, Converti RM. Postural disorders in conservatory students: the Diesis project. Med Probl Perform Art. 2014 Mar;29(1):19-22. doi: 10.21091/mppa.2014.1005. PMID 24647457
- [Background] undefined
- [Background] Steinmetz A, Scheffer I, Esmer E, Delank KS, Peroz I. Frequency, severity and predictors of playing-related musculoskeletal pain in professional orchestral musicians in Germany. Clin Rheumatol. 2015 May;34(5):965-73. doi: 10.1007/s10067-013-2470-5. Epub 2014 Jan 5. PMID 24389813
- [Background] Kok LM, Huisstede BM, Voorn VM, Schoones JW, Nelissen RG. The occurrence of musculoskeletal complaints among professional musicians: a systematic review. Int Arch Occup Environ Health. 2016 Apr;89(3):373-96. doi: 10.1007/s00420-015-1090-6. Epub 2015 Nov 12. PMID 26563718
- [Background] Cruder C, Barbero M, Koufaki P, Soldini E, Gleeson N. Prevalence and associated factors of playing-related musculoskeletal disorders among music students in Europe. Baseline findings from the Risk of Music Students (RISMUS) longitudinal multicentre study. PLoS One. 2020 Dec 9;15(12):e0242660. doi: 10.1371/journal.pone.0242660. eCollection 2020. PMID 33296381
- [Background] Zaza C, Charles C, Muszynski A. The meaning of playing-related musculoskeletal disorders to classical musicians. Soc Sci Med. 1998 Dec;47(12):2013-23. doi: 10.1016/s0277-9536(98)00307-4. PMID 10075243